CLINICAL TRIAL: NCT05532228
Title: Evaluation of the Functional Impact of Adenotonsilectomy in Children
Brief Title: Evaluation of the Functional Impact of Adenotonsilectomy
Status: Completed | Type: Observational
Sponsor: Instituto de Ciências Biomédicas Abel Salazar (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.176(137-DEFI/139-CE)
Record Dates: First submitted 2022-07-14; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Apnea, Obstructive; Tonsillitis; Tonsillar Hypertrophy; Respiratory Function Impaired; Infections; ENT Disorder
Keywords: adenotonsillectomy; children; spirometry; obstructive sleep apnea; adenotonsillar hypertrophy; respiratory function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis; Respiratory Insufficiency; Infections; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obstructive sleep apnea: children with adenotonsillar hypertrophy and reports of nocturnal arousals/gasp/respiratory abnormalities
  Interventions: Procedure: Adenotonsillectomy
- No obstructive sleep apnea: children without adenotonsillar hypertrophy and no reports of nocturnal arousals/gasp/respiratory abnormalities
  Interventions: Procedure: Adenotonsillectomy
- Recurrent infections: Children with recurrent upper respiratory infections
  Interventions: Procedure: Adenotonsillectomy
- no recurrent infections: Children without recurrent upper respiratory infections
  Interventions: Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: Adenotonsillectomy — adenotonsillectomy by cold dissection

SUMMARY:
Spirometric assessment of respiratory function before and after adenotonsillectomy surgery

DETAILED DESCRIPTION:
Spirometric assessment of respiratory function before and after adenotonsillectomy surgery Study site at CHUPorto: Department of Otorhinolaryngology at CHUPorto, Portugal.

Study design: Institutional, observational, cohort, prospective. Classification of studies according to the law of clinical investigation (Dec. Law No. 21/2014): Clinical study without intervention. Main objective of the study: To collect a database referring to pediatric patients enrolled for surgery in an outpatient setting, in order to compare vital, spirometric and clinical parameters at two different times: pre and post surgical intervention.

Secondary objectives of the study: Based on validated indices, to assess the impact of surgical intervention on the child's respiratory and cardiovascular system. Participants: Patients undergoing surgery in the field of Pediatric Otorhinolaryngology at CHUPorto, a tertiary referral Hospital in Portugal.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4-14 years;
* Patients with surgical indication for any combination of:

  * tonsillectomy
  * adenoidectomy
  * turbinoplasty
  * myringotomy;
* naive children (not submitted to previous ENT surgery);
* signature of informed consent by the parent entity.

Exclusion Criteria:

* Age under 4 years and over 14 years;
* surgery: myringotomy+TT placement exclusively;
* associated co-morbidities:

  * asthma/other obstructive lung diseases
  * congenital facial or thoracic dysmorphism
  * neurological disease with cognitive impairment
  * cardiopulmonary disease
* patients without surgical indication
* other causes of nasal obstruction (severe septum deviation or polyps).

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing surgery within the scope of Pediatric Otorhinolaryngology at CHUPorto.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in the first second (FEV 1) | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
Forced vital capacity (FVC) | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
Peak expiratory flow (PEF) | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
forced expiratory flow rate at 25% (F25) | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
forced expiratory flow rate at 75% (F75) | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
forced expiratory flow between 25 and 75% of the pulmonary volume (FEF25-75%). | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.

SECONDARY OUTCOMES:
Weight | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
Diastolic arterial pressure | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
Systolic arterial pressure | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
Heart rate | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery.
rest oxygen saturation | 3 months after surgery
  Measured in two moments by the same operator: pre-operatively, in the day of intervention and post-operatively, 3 months after surgery. (through instant photoplethysmography in the index finger with the patient in a calm environment

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Univrsitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data